CLINICAL TRIAL: NCT02099409
Title: Open Label Single Center Randomized Cross Over Study to Validate Current Algorithms and Evaluate Safety and Efficacy of Closed Loop Insulin Delivery (FlorenceD2 System) in Children With Type 1 Diabetes Between 6 - 12 Years of Age
Brief Title: Safety and Efficacy of Overnight Closed Loop in Children With Type 1Diabetes Mellitus in Luxembourg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier du Luxembourg (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, Carine de Beaufort, MD , PhD, Centre Hospitalier du Luxembourg
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SPIDLUX 4
Record Dates: First submitted 2014-03-26; First posted 2014-03-28 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 diabetes mellitus; children; closed loop; cross over; overnight; FLORENCED2; DANA Diabecare R pump; FreeStyle Navigator II; Dexcom G4
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Starting with FLORENCED2 followed by open loop (Experimental): Start 2 Overnight periods with closed loop through FLORENCED2 Device , followed by 2 overnight periods with open loop.
  Interventions: Device: FLORENCED2
- Start open loop followed by FLORENCED2 (Experimental): Start with 2 overnight periods with open loop , followed by 2 overnight with closed loop FLORENCED2
  Interventions: Device: FLORENCED2

INTERVENTIONS:
Device: FLORENCED2 — FLORENCED2 device ensures the closed loop between Freestyle Navigator II and the DANA DIABECARE R

SUMMARY:
The purpose of this study is to validate current algorithms and evaluate safety and efficacy of overnight closed loop insulin delivery (FlorenceD2 system) in children with type 1 diabetes between 6 - 12 years of age in Luxembourg .

ELIGIBILITY:
Inclusion Criteria:

* Between 6 - ≤12 years
* With type 1 diabetes for 6 months or more and
* Pump user for at least 6 months.
* HbAc1 should be <11 %.
* No medication or physical or psychological disease should be present, which could interfere with the study.

Exclusion Criteria:

-None

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Time spent in normal glucose range ( mg/dl) | At least 5 hours between 7 pm and 7 am
  Glucose will be measured with a Continuous glucose monitoring device

SECONDARY OUTCOMES:
glucose variability ( excursions in mg/dl) | 7 pm - 7 am
  Continuous Glucose Monitoring device
Time spent in low glucose range (< 60 mg/dl) | 7 pm till 7 am
  Continuous Glucose Monitoring
time spent in low glucose range (<70 mg/dl) | 7 pm till 7 am
  continuous glucose monitoring
time spent in high glucose range (>180mg/dl) | 7 pm - 7 am
  continuous glucose monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Carine deBeaufort, MD PhD, Principal Investigator — Centre Hospitalier du Luxembourg; Roman Hovorka, Professor, Principal Investigator — University of Cambridge; Gosia Wilinska, PhD, Principal Investigator — University of Cambridge; Ulrike Schierloh, MD, Principal Investigator — Centre Hospitalier du Luxembourg
Locations (2):
- Luxembourg (2):
  - DECCP Clinique Pédiatrique de Luxembourg/CHL, Luxembourg
  - DECCP Pediatric Clinic , CHLuxembourg, Luxembourg